CLINICAL TRIAL: NCT06000644
Title: Effects of Progressive Combined Cognitive Training and Rhythmic Auditory Stimulation in Treadmill Training on Walking Automaticity, Executive Function, and Dual-task Coordination for Patients With Chronic Stroke
Brief Title: Effects of Combined Cognitive Training and Rhythmic Auditory Stimulation in Treadmill Training After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Li-Ling Chuang, Associated Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPD1M0841
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: stroke; gait rehabilitation; rhythmic auditory stimulation; cognitive training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- combined group (Experimental): The combined group will undertake progressive treadmill walking speed while performing a cognitive task with rhythmic auditory cueing.
  Interventions: Device: Combined group
- cognitive group (Active Comparator): The cognitive group will receive cognitive training while walking on the treadmill.
  Interventions: Device: Cognitive group
- rhythmic group (Active Comparator): The rhythmic group will hear rhythmic auditory stimulation while treadmill walking.
  Interventions: Device: Rhythmic group
- treadmill group (Active Comparator): The treadmill group will train only in progressive treadmill walking.
  Interventions: Device: Treadmill group

INTERVENTIONS:
Device: Combined group — The combined group will undertake progressive treadmill walking speed while performing a cognitive task with rhythmic auditory cueing for 30 minutes per session, 3 times a week for 4 weeks.
  Arms: combined group
Device: Cognitive group — The cognitive group will receive cognitive training while treadmill walking with a progressive speed for 30 minutes per session, 3 times a week for 4 weeks .
  Arms: cognitive group
Device: Rhythmic group — The rhythmic group will hear rhythmic auditory stimulation while treadmill walking for 30 minutes per session, 3 times a week for 4 weeks.
  Arms: rhythmic group
Device: Treadmill group — The treadmill group will train only in progressive treadmill walking for 30 minutes per session, 3 times a week for 4 weeks.
  Arms: treadmill group

SUMMARY:
The objective of this study is to compare the effects of progressive combined cognitive training and rhythmic auditory stimulation to treadmill training (combined group), cognitive treadmill training (cognitive group), rhythmic auditory stimulation to treadmill training (rhythmic group), and treadmill walking alone (treadmill group) on walking automaticity, executive function, and dual-task coordination for patients with chronic stroke (Aim 1). The second aim of this study is to investigate the factors affecting the results of interventions (Aim 2). The third aim of the study is to examine the characteristics of stroke population who are appropriate for progressive combined cognitive training and rhythmic auditory stimulation to treadmill training.

DETAILED DESCRIPTION:
A single-blinded, randomized controlled trial will be conducted at medical centers. Eighty stroke patients will be randomized to one of the four groups. All groups will receive interventions 30 minutes per time, 3 times a week, for 4 weeks. The combined group will undertake progressive treadmill walking speed and rhythmic auditory stimulation while performing a cognitive task. The cognitive group will receive cognitive training while walking on the treadmill. The rhythmic group will hear rhythmic auditory stimulation while treadmill walking. The treadmill group will train only in progressive treadmill walking. A blinded assessor will administer three assessments. All participants will be examined for gait and cognitive performance under single-task (walking only, Stroop task only) and dual-task conditions (walking while performing the Stroop task) at baseline, post-intervention, and one-month follow-up. The primary outcome measures of gait and cognition are gait speed and cognitive score of the Stroop task under single- and dual-task conditions. The secondary outcome measures are the Mini-BESTest, Walking Ability Questionnaire, 6-minute Walk Test, and Stroke Impact Scale. Repeated measure ANOVA will be used to compare measurements at baseline, after training, and follow-up between and within the groups.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with first-time stroke;
2. more than 6 months after stroke onset;
3. able to walk 10 meters;
4. no severe vision, hearing, or speech impairments;
5. understand and follow the instructions and sign the Informed Consent Form;
6. older than 20 years old.

Exclusion Criteria:

1. orthopedic problems affecting walking or other diseases that may interfere with study participation;
2. a score of less than 24 on the mini-mental state examination (MMSE);
3. severe balance disorder with a total score of less than 45 points Berg Balance Scale.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Walking speed (m/s) | 5 minutes
  Participants will walk 10 meters at their preferred speed with and without the Stroop task twice, respectively. The spatiotemporal gait parameters will be examined using Physilog® sensors (Gait Up, Switzerland) and analyzed by the Gait Analysis Package software on the USB key. Walking speed (m/s) is the mean speed of forward walking, calculated in meters per second.
Stride time variability (%) | 5 minutes
  The stride time is the duration of one cycle (from heel strike to heel strike of the same side). Stride time variability (%) is the coefficient of variation of stride time or cycle duration in percent.
Gait asymmetry (%) | 5 minutes
  Gait asymmetry will be assessed by comparing left and right swing time, in percent. A perfect symmetry outputs a value of 0%.
Cognitive composite score | 5 minutes
  The Stroop task is the commonly utilized dual-task paradigm and measures executive function and response inhibition, which plays a vital role during walking. Therefore, the Stroop task will be selected to assess cognitive dual-task walking. The Stroop task will be performed while sitting and walking to assess executive function under single-task and dual-task conditions. The following is the formula for calculating the cognitive composite score: Cognitive composite score of the Stroop task = [Accuracy(%)/Reaction time(milliseconds)] * 100. The better the cognitive performance of the Stroop task, the higher the cognitive composite score.
  The instructions for the dual-task walking (walking + Stroop) are designed to encourage neutral prioritization between the two tasks ("walk at the preferred speed while performing the Stroop task as accurately and quickly as you can").

SECONDARY OUTCOMES:
Dual-task automaticity | 5 minutes
  Automaticity is based on the combined interference of both motor (i.e., walking speed) and cognitive DTE. The combined dual-task effect (cDTE) is a measure that quantifies automaticity while performing a dual-task. The walking speed and cognitive composite score under single-task and dual-task conditions will be used to calculate combined DTE.A negative cDTE value is indicative of automaticity under dual-task that deteriorated or interfered. A positive cDTE value indicates automaticity facilitation.
Task-specific dual-task interference | 5 minutes
  Task-specific dual-task interference calculates the motor (i.e., walking speed) or cognitive dual-task effect (DTE), which relates dual-task performance to single-task performance. For assessing dual-task interference, quantifying the combined interference of the motor and the cognitive tasks may be a more comprehensive measure of the dual-task effect to provide a more accurate picture of gait automaticity. The walking speed and cognitive composite score will be used to calculate motor and cognitive dual-task effect (DTE). For both the motor (i.e., walking speed) and cognitive DTE in this study, negative DTE values (i.e., dual-task interfence) indicate poor performance under dual-task walking condition compared to single-task conditions.
6-minute Walking test, 6MWT | 6 minutes
  The 6-minute walk test will be used to measure participants' walking capacity and walking endurance.The participants will ask to walk for six minutes at their own pace, resting or slowing down as needed, and the total distance (meters) of walking in six minutes will be recorded
Stroke impact scale, SIS | 10 minutes
  The SIS was developed to measure the quality of life after a stroke. The SIS 3.0 has eight domains: strength, hand function, mobility, activities of daily living/instrumental activities of daily living (i.e., ADLs and IADLs), memory and thinking, communication, emotion, and social participation. Scores for each domain range from 0 to 100, and higher scores indicate a better health-related quality of life. Lower scores indicate more incredible difficulty in task completion during the past week or past two weeks, or past four weeks. Eight items on the social participation domain and eight items on the mobility domain of the SIS will be used to measure the social participation of individuals with chronic stroke in this study.
Mini-Balance Evaluation System Test, Mini-BESTest | 10 minutes
  The Mini-BESTest is a reliable and valid tool for evaluating balance in people with chronic stroke. It consists of 14 items and includes four subscales: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Each test item is rated on a three-point ordinal scale (0-2, 0=severe, 1=moderate, and 2=normal), with the total score ranging between 0 and 28 points.
Walking ability questionnaire | 5 minutes
  The walking ability questionnaire was designed to provide a more detailed assessment of the individual's social limitations due to reduced walking ability. A research assistant will administer the questionnaire to rate the participant's current customary mobility of 19 ambulatory activities performed in the home (8 items) and community (11 items). Current customary mobility was defined as an individual's self-reported ability to enter and leave the listed locations. Each test item is rated on a five-point ordinal scale (0-4, 0= unable, 1= wheelchair, 2="assisted, 3= supervised, 4= independent). An overall score was calculated. The range of scale was 0 to 76.
Outdoor walking assessment | 15 minutes
  Participants will walk 400 meters at their comfortable speed on the street. A 402-meter walkway will be used for outdoor walking test. In order to allow the participants to have enough distance to accelerate and decelerate, only the time taken the middle 400 meters will be recorded by a stopwatch. The outcome measure will be walking speed (m/s).

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ling Chuang, Ph.D., Principal Investigator — Chang Gung University
Locations (1):
- Mackay Memory Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No